CLINICAL TRIAL: NCT07075003
Title: Effect of NOL-Guided vs Conventional Intraoperative Opioid Infusion on Outcomes in Geriatric Patients Undergoing Lumbar Stabilization Surgery
Brief Title: NOL-Guided vs Conventional Intraoperative Opioid Infusion on Outcomes in Geriatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Süheyla Abitağaoğlu, Associate Professor, MD, Saglik Bilimleri Universitesi
Other Study IDs: sabitagaoglu
Record Dates: First submitted 2025-07-01; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Pain; Opioid Use; Geriatric Anesthesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conservative: Our clinic's standard anesthesia induction and maintenance method will be applied to all patients. Patients will receive standard monitoring including peripheral oxygen saturation, non-invasive blood pressure, ECG, and anesthesia depth. All patients will receive intravenous 2-2.5 mg/kg propofol under Sedline guidance, and remifentanil via target-controlled infusion at an effect-site concentration of 4 ng/ml. After anesthesia depth falls below 50, 0.6 mg/kg rocuronium will be administered. Maintenance anesthesia will be with 1-2% sevoflurane in 40/60% oxygen/air mixture at 2 L flow.Remifentanil is administered as a continuous infusion in conservative approach;dosage adjustments are made based on heart rate and blood pressure changes to estimate pain levels.
- Nociceptive level: Our clinic's standard anesthesia induction and maintenance method will be applied to all patients. Patients will receive standard monitoring including peripheral oxygen saturation, non-invasive blood pressure, ECG, and anesthesia depth. All patients will receive intravenous 2-2.5 mg/kg propofol under Sedline guidance, and remifentanil via target-controlled infusion at an effect-site concentration of 4 ng/ml. After anesthesia depth falls below 50, 0.6 mg/kg rocuronium will be administered. Maintenance anesthesia will be with 1-2% sevoflurane in 40/60% oxygen/air mixture at 2 L flow.Remifentanil is administered as a continuous infusion by using Nociceptive level guidance
  Interventions: Device: nociceptive level

INTERVENTIONS:
Device: nociceptive level — remifentanil infusion dose adjustment according to the changes of nociceptive level
  Groups: Nociceptive level

SUMMARY:
The aim of this study is to compare the effects of conventional methods and goal-directed therapy guided by pain monitoring on total remifentanil dosage, wake-up time, and complications in geriatric patients undergoing lumbar stabilization surgery.

DETAILED DESCRIPTION:
With the aging population, the number of geriatric patients undergoing surgery is increasing daily. One of the anesthesiologists' main responsibilities is to prevent intraoperative pain and related complications. Opioids have been known for thousands of years as valuable tools for pain management and remain the cornerstone of perioperative analgesia today (1). Remifentanil is currently the most commonly used opioid during the intraoperative period due to its potent analgesic properties, short duration of action, and metabolism by plasma enzymes. While it may improve hemodynamic stability, remifentanil can also cause hypotension and bradycardia. Prolonged remifentanil use may lead to hyperalgesia, increasing the need for postoperative opioid analgesics and consequently leading to opioid-related side effects. In elderly patients, changes in body composition, drug sensitivity, and hepatic/renal metabolism require more cautious opioid administration.

Optimizing remifentanil infusion dosing during surgery may reduce total opioid consumption and thus decrease side effects such as wake-up time, postoperative pain, and nausea.

In conventional use, remifentanil is administered as a continuous infusion, and dosage adjustments are made based on heart rate and blood pressure changes to estimate pain levels. However, with goal-directed therapy guided by pain monitoring, more effective analgesia can be achieved. These applications are selected based on the clinician's experience and preferences. While some publications report that total remifentanil use decreases in patients with dose adjustments guided by pain monitoring, evidence is lacking regarding which method is superior in terms of patient outcomes in elderly populations.The aim of this study is to compare the effects of conventional methods and goal-directed therapy guided by pain monitoring on total remifentanil dosage, wake-up time, and complications in geriatric patients undergoing lumbar stabilization surgery.

After obtaining informed consent, a total of 80 geriatric patients undergoing lumbar stabilization surgery will be included. Once on the operating table, all patients will receive standard monitoring including peripheral oxygen saturation, non-invasive blood pressure, ECG, and anesthesia depth. All patients will receive intravenous 2-2.5 mg/kg propofol under Sedline guidance, and remifentanil via target-controlled infusion at an effect-site concentration of 4 ng/ml. After anesthesia depth falls below 50, 0.6 mg/kg rocuronium will be administered. Maintenance anesthesia will be with 1-2% sevoflurane in 40/60% oxygen/air mixture at 2 L flow. The method of remifentanil administration will be determined by the attending anesthesiologist.

Demographic data (age, height, weight, gender, comorbidities, ASA score) will be recorded. Hemodynamic parameters (blood pressure, heart rate, oxygen saturation, end-tidal CO₂), remifentanil dosage, and NOL levels (for Group 2) will be recorded every 15 minutes during the surgery. At the end of surgery, the following will be documented:

Total remifentanil dosage Blood loss and transfusion volume Number of hypotensive events (MAP <55) Wake-up time Total surgical time NRS (Numerical Rating Scale) pain scores Nausea-vomiting scores

In the post-anesthesia care unit (PACU), pain and nausea-vomiting scores will be evaluated at the 10th, 20th, and 30th minutes, along with duration of PACU stay. During ward follow-up, pain scores, nausea-vomiting scores, administered medications, and length of postoperative hospital stay will be recorded at 1, 3, 6, and 24 hours.

Nausea-vomiting will be assessed using a 4-point scale:

0: none

1. nausea without vomiting
2. nausea with vomiting
3. vomiting more than twice

Pain will be assessed using the NRS scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar stabilization surgery

Exclusion Criteria:

* Chronic opioid use
* Severe congestive heart failıure
* Severe arrhythmia
* Uncontrolled hypertension

Ages: 65 Years to 90 Years | Sex: All
Age Groups: Older Adult
Study Population: A total of 80 geriatric patients undergoing lumbar stabilization surgery
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Total dose | operation duration
  Total dose of remifentanil used in operation

SECONDARY OUTCOMES:
postoperative pain | postoperative 10th, 20th, and 30th minutes, 1, 3, 6, and 24 hours
  pain evaluation during postoperative 24 hour,
  11 point Numeric Rating Scale (NRS) will be used to measure pain level (0-10) 0: No pain, 10: Worst possible pain
nausea and vomiting | postoperative 10th, 20th, and 30th minutes, 1, 3, 6, and 24 hours
  postoperative nausea and vomiting
  Nausea-vomiting will be assessed using a 4-point scale:
  0: none
  1. nausea without vomiting
  2. nausea with vomiting
  3. vomiting more than twice

CONTACTS AND LOCATIONS:
Overall Officials: Süheyla Abitağaoğlu, Principal Investigator — UNIVERSİTY OF HEALTH SCIENCES

REFERENCES:
- [Background] Gazelka HM, Leal JC, Lapid MI, Rummans TA. Opioids in Older Adults: Indications, Prescribing, Complications, and Alternative Therapies for Primary Care. Mayo Clin Proc. 2020 Apr;95(4):793-800. doi: 10.1016/j.mayocp.2020.02.002. PMID 32247352
- [Background] Hwang W, Lee J, Park J, Joo J. Dexmedetomidine versus remifentanil in postoperative pain control after spinal surgery: a randomized controlled study. BMC Anesthesiol. 2015 Feb 24;15:21. doi: 10.1186/s12871-015-0004-1. eCollection 2015. PMID 25750586
- [Background] Mercadante S. Influence of aging on opioid dosing for perioperative pain management: a focus on pharmacokinetics. J Anesth Analg Crit Care. 2024 Aug 1;4(1):51. doi: 10.1186/s44158-024-00182-2. PMID 39085914